CLINICAL TRIAL: NCT00972309
Title: A Pilot Study of Vaccination With Epitope-Enhanced TARP Peptide and TARP Peptide-Pulsed Dendritic Cells in the Treatment of Stage D0 Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090139; 09-C-0139; NCT00908258 (obsolete NCT alias)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Prostate Specific Antigens; Prostate Neoplasms
Keywords: Epitope-Enhanced TARP Peptide; Prostate Cancer; TARP Peptide-Pulsed Dendritic Cells; PSADT; HLA-A*0201
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TARP; Protein Subunit Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: T-cell receptor alternate reading frame protein (TARP) (Experimental): TARP peptides
  Interventions: Biological: T-cell receptor alternate reading frame protein (TARP) peptide vaccine
- Cohort: 2 -T-cell receptor alternate reading frame protein (TARP) (Experimental): TARP dendritic cells
  Interventions: Biological: T-cell receptor alternate reading frame protein (TARP) dendritic cell vaccine

INTERVENTIONS:
Biological: T-cell receptor alternate reading frame protein (TARP) peptide vaccine — Will receive an admixture of the wildtype and epitope enhanced TARP peptides emulsified with Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF). TARP peptide will be administered subcutaneously at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96
  Arms: Cohort 1: T-cell receptor alternate reading frame protein (TARP)
Biological: T-cell receptor alternate reading frame protein (TARP) dendritic cell vaccine — Will receive peptide pulsed dendritic cells administered intradermally in two vaccination sites. TARP pulsed dendritic cells will be administered at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.
  Arms: Cohort: 2 -T-cell receptor alternate reading frame protein (TARP)

SUMMARY:
Background:

* PSA (prostate specific antigen) is a protein found on normal and cancerous prostate cells. Levels of this protein are used to identify men who are at risk for prostate cancer and to monitor responses to treatment in men who have been diagnosed with prostate cancer.
* Research has shown that men who continue to have an elevated PSA level following primary treatment for prostate cancer are at increased risk for cancer progression. Studies have shown that the change in PSA levels over time, or PSA doubling time (PSADT), can be accurate in predicting how quickly the cancer is likely to progress. Individuals with a PSADT of less than 3 months are at extremely high risk for disease progression and death from prostate cancer. Individuals with a PSADT of greater than 15 months have a very low risk of death from prostate cancer.
* T-cell receptor alternate reading frame protein (TARP) is a protein that is found in about 95% of prostate cancers and is known to stimulate the immune system. The TARP prostate cancer vaccine is made from pieces of the TARP protein called peptides and includes peptides that have been modified to make them more effective at stimulating immunity. Although these TARP peptides have been shown to stimulate the immune systems of mice, information is needed to determine if they also stimulate the immune system in humans. Since it is unclear what is the best way to give peptide vaccines, the TARP peptides will be given with substances known to stimulate the immune system or in a vaccine made with the patient s own cells.

Objectives:

* To determine the immune systems response to vaccination with TARP peptides.
* To determine the safety and toxicity of TARP peptide vaccination.
* To determine if vaccination with the TARP prostate cancer vaccine can slow down PSADT in men with an intermediate PSADT of 3 to 15 months.

Eligibility:

* Males 18 years of age and older who have completed their primary treatment for prostate cancer, have stage D0 disease, are Human leukocyte antigen (HLA) A*0201 positive and who have a PSADT greater than 3 and less than 15 months.

Design:

* Patients will be randomized to one of two treatment arms:
* Arm A will receive the TARP vaccine with other substances that stimulate the immune system.
* Arm B will receive the TARP vaccine that includes a patients own white blood cells.
* First week of study, after screening for eligibility has been completed:
* Day 1: Apheresis procedure to extract white blood cells to test the immune response to the vaccine.
* Day 3: Flu vaccine to allow researchers to determine how well a patients immune system is working.
* Clinic visits in Weeks 3, 6, 9, 12, and 15 for physical examination, blood samples, and administration of the TARP peptide vaccine.
* Physical examination and blood samples only in Weeks 18 and 36.
* Additional blood samples and apheresis procedures in Weeks 24 and 48.
* A 6th dose of TARP peptide vaccine will be administer to those patients who have a response to vaccination at week 24.
* No follow-up or long-term study is associated with this study.

DETAILED DESCRIPTION:
BACKGROUND:

* T-cell receptor alternate reading frame protein (TARP) is expressed by both normal and malignant prostate cancer tissue and is found in about 95% of prostate cancer specimens. TARP is immunogenic and hence is a target antigen for vaccination.
* The immunogenicity of TARP peptides can be augmented through epitope enhancement that is achieved through amino acid substitutions resulting in increased peptide binding affinity.
* Two HLA-A*0201 TARP peptide epitopes are associated with generation of catalytic T-cell responses: TARP27-35 and TARP29-37. Substitution of Val for Leu at position 9 in TARP29-37, results in a peptide with increased binding affinity (TARP29-37-9V) that induces antigen specific T cells able to recognize wild type and multiple modified TARP peptides. The affinity of the TARP 27-35 peptide, corresponding to a distinct but overlapping epitope, is high enough that no enhancement was required.
* Stage D0 prostate cancer patients have no evidence of visceral or bony metastatic disease but have persistently elevated or rising prostate-specific antigen (PSA) levels (biochemical progression) and are at increased risk for disease progression. Since they lack much of the immune dysfunction associated with the high tumor burden characteristic of end-stage metastatic disease, they are an ideal population in which to study therapeutic vaccination to slow or prevent disease recurrence and progression.
* Dendritic cells (DC) are the most potent antigen-presenting cells of the immune system and are being studied extensively for anti-tumor activity in a broad spectrum of cancer patients.
* As the optimal method for therapeutic immunization with peptide vaccines in patients with cancer is unclear, vaccination with TARP peptides in Montanide ISA 51 VG adjuvant plus Sargramostim will be studied in a randomized fashion with autologous, TARP peptide-pulsed dendritic cells (DCs) in HLA-A*0201 Stage D0 prostate cancer patients.

OBJECTIVES:

* Determine the safety and toxicity of TARP peptide and TARP peptide-pulsed dendritic cell vaccination in patients with Stage D0 prostate cancer.
* Determine the T-lymphocyte immune responses to TARP peptide vaccination with Montanide ISA 51 VG plus Sargramostim or autologous dendritic cells as measured by tetramer staining, interferon (IFN)-gamma enzyme-linked immune absorbent spot (ELISpot) and (51)Cr release cytotoxic T lymphocytes (CTL) assays.

ELIGIBILITY:

* Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate.
* Must have completed and recovered from all prior definitive therapy (surgery, brachytherapy, cryotherapy or radiotherapy) for the primary tumor, or other definitive-intent local therapy.
* Stage D0 disease with documented biochemical progression documented by rising PSA and no evidence of metastatic disease by physical examination, computed tomography (CT) scan or bone scan.
* Prostate-specific antigen doubling time (PSADT) greater than or equal to 3 months and less than or equal to or equal to 15 months:

  * Patients must have greater than or equal to 3 PSA measurements over greater than or equal to 3 months.
  * The interval between PSA measurements must be greater than or equal to 4 weeks.
* For patients following definitive radiation therapy or cryotherapy: a rise in PSA of > 2ng/mL above the nadir (per Radiation Therapy Oncology Group (RTOG)-American Society for Radiation Oncology (ASSTRO) consensus criteria).
* For patients following radical prostatectomy: 2 absolute PSA values > 0.3ng/ml (per National Comprehensive Cancer Network (NCCN) guidelines).
* Non-castrate level of testosterone: greater than or equal to 50 ng/dL (prior androgen deprivation therapy (ADT) allowed; must be greater than or equal to 6 months since last dose of ADT).
* HLA-A*0201 positive.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-2 or Karnofsky 70-100% and life expectancy greater than or equal to 1 year.
* Hemoglobin greater than or equal to 10.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500/mm(3), absolute lymphocyte count (ALC) greater than or equal to 500/ mm(3), absolute neutrophil count (ANC) greater than or equal to 1,000/mm(3), platelet count greater than or equal to 100,000/mm(3), and prothrombin time (PT)/partial thromboplastin time (PTT) less than or equal to 1.5 times upper limits of normal (ULN) unless receiving clinically indicated anticoagulant therapy; serum glutamic pyruvic transaminase (SGPT)/Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 times ULN, total bilirubin less than or equal to 1.5 times ULN; creatinine less than or equal to 1.5 times ULN and estimated glomerular filtration rate (GFR) estimated glomerular filtration rate (eGFR) greater than or equal to 60 ml/min.
* Hepatitis B and C negative (unless the result is consistent with prior vaccination or prior infection with full recovery); human immunodeficiency virus (HIV) negative.
* No use of investigational agents within 4 weeks of study enrollment or use of immunosuppressive or immunomodulating agents within 8 weeks of study entry.
* No other concurrent anticancer therapy or prior prostate cancer vaccines expressing TARP or human leukocyte antigen (HLA) A2.
* No alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto). Note: patients receiving medications for urinary symptoms such as Flomax or 5-alpha reductase inhibitors (finasteride and dutasteride) on a chronic stable dose for at least 3 months are allowed.

STUDY DESIGN:

* This is a randomized, prospective, pilot study of vaccination with a mixture of wild type (TARP27-35) and epitope-enhanced (TARP29-37-9V) TARP peptides in HLA-A*0201 patients with stage D0 prostate cancer.
* Vaccination with TARP peptides admixed with Montanide ISA 51 VG plus Sargramostim administered by deep subcutaneous injection will be compared with vaccination with TARP peptide-pulsed autologous dendritic cells (DCs) administered intradermally.
* Autologous dendritic cells will be matured from peripheral blood monocytes with Sargramostim, interleukin 4 (IL4), IFN-gamma and LPS and pulsed with wild type and epitope-enhanced TARP peptides.
* Apheresis will be performed on all patients at weeks 0, 24, 48 and 96.
* Randomization and assignment to received TARP peptide vaccine with Montanide ISA 51 VG plus Sargramostim given by deep subcutaneous injection or TARP peptide-pulsed autologous DCs given ID will be performed at week 0.
* All patients will receive live, attenuated influenza vaccine (FluMist) when seasonally available at the very end of their week 0 visit as a control vaccine to assess cytotoxic T lymphocyte responses.
* TARP Peptide vaccines will be administered every three weeks at weeks 3, 6, 9, 12, and 15, with a sixth and seventh booster dose of vaccine at Week 48 and 96. Follow-up will be through 144 weeks on study.
* The trial uses an optimal 2-stage design targeting an immunologic response between 10 and 40%. We will initially accrue 9 patients in each arm. If 0-1 patients develop an immunologic response, then no further patients will be enrolled. If 2 or more of these patients develop an immunologic response, we will accrue 11 additional patients for a maximum total of up to 20 patients in each arm. A stopping rule for excessive toxicity will be incorporated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate.
* Human leukocyte antigen-A (HLA-A)*201 positive
* Patients must have
* Completed and recovered from all prior definitive therapy (surgery, brachytherapy, cryotherapy or radiotherapy) for the primary tumor, or other definitive-intent local therapy.
* Stage D0 disease with documented biochemical progression documented by a rising prostate-specific antigen (PSA).
* No evidence of metastatic disease by physical examination, computed tomography (CT) scan or bone scan.
* For patients following definitive radiation therapy or cryotherapy: a rise in PSA of >2ng/mL above the nadir.
* For patients following radical prostatectomy: 2 absolute PSA values > 0.3 ng/mL
* Non-castrate level of testosterone: greater than or equal to 50 ng/dL (prior androgen deprivation treatment (ADT) allowed; must be greater than or equal to 6 months since last dose of ADT).
* A Pre-Enrollment/Baseline prostate-specific antigen doubling time (PSADT) > 3 months and less than or equal to 15 months
* Patients must have greater than or equal to 3 PSA measurements over greater than or equal to 3 months
* The interval between PSA measurements must be greater than or equal to 4 weeks
* For patients receiving 5-alpha reductase inhibitors (5ARI) e.g. finasteride or dutasteride, only PSA values obtained after at least 3 months on therapy may be used to calculate PSADT.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-2 or Karnofsky 70-100%
* Life expectancy greater than or equal to 1 year.
* Hemoglobin greater than or equal to 10.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500/mm(3), absolute lymphocyte count (ALC) greater than or equal to 500/mm(3), absolute neutrophil count (ANC) greater than or equal to 1,000/mm(3), platelet count greater than or equal to 100,000/mm(3).
* Prothrombin time (PT)/ partial thromboplastin time (PTT) less than or equal to 1.5 times upper limits of normal (ULN) unless receiving clinically indicated anticoagulant therapy.
* Serum glutamic oxaloacetic transaminase (SGOT)/Serum glutamic pyruvic transaminase (SGPT) < 2.5 times ULN, total bilirubin < 1.5 times ULN, creatinine (Cr) < 1.5 times ULN, estimated glomerular filtration rate (GFR) estimated glomerular filtration rate (eGFR) > 60 ml/min.
* Hepatitis B and C negative, unless the result is consistent with prior vaccination or prior infection with full recovery.
* Human immunodeficiency virus (HIV) negative
* No use of investigational agents within 4 weeks of study enrollment.
* No use of immunosuppressive (cytotoxic chemotherapy, systemic steroids) or immunomodulating agents (including intravenous immune globulin (IVIG) within 8 weeks of study entry. Note: topical and intranasal steroid therapy is permitted.
* No other concurrent anticancer therapy.
* No alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto). Note: patients receiving medications for urinary symptoms such as Flomax or 5-alpha reductase inhibitors (finasteride and dutasteride) on a chronic stable dose for at least 3 months are allowed.
* No prior prostate cancer vaccines expressing TARP or HLA A2.
* Able to understand and provide Informed Consent.

EXCLUSION CRITERIA:

* HLA-A*201 negative
* Patients with an active second malignancy other than adequately treated squamous or basal cell carcinoma of the skin, or superficial bladder carcinoma.
* Patients with active infection.
* Patients with brain, visceral or bony metastatic disease.
* Patients in who live attenuated intranasal influenza vaccine (FluMist) is contraindicated including individuals with asthma or reactive airways disease, cardiovascular or pulmonary disease, chronic metabolic diseases (including diabetes mellitus), renal dysfunction or hemoglobinopathies.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-05-11 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Stern LJ, Wiley DC. Antigenic peptide binding by class I and class II histocompatibility proteins. Behring Inst Mitt. 1994 Jul;(94):1-10. No abstract available. PMID 7998902
- [Background] Berzofsky JA, Ahlers JD, Belyakov IM. Strategies for designing and optimizing new generation vaccines. Nat Rev Immunol. 2001 Dec;1(3):209-19. doi: 10.1038/35105075. PMID 11905830
- [Background] Rivoltini L, Squarcina P, Loftus DJ, Castelli C, Tarsini P, Mazzocchi A, Rini F, Viggiano V, Belli F, Parmiani G. A superagonist variant of peptide MART1/Melan A27-35 elicits anti-melanoma CD8+ T cells with enhanced functional characteristics: implication for more effective immunotherapy. Cancer Res. 1999 Jan 15;59(2):301-6. PMID 9927036
- [Derived] Berzofsky JA, Wood LV, Terabe M. Cancer vaccines: 21st century approaches to harnessing an ancient modality to fight cancer. Expert Rev Vaccines. 2013 Oct;12(10):1115-8. doi: 10.1586/14760584.2013.836906. No abstract available. PMID 24124874
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0139.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF): T-cell receptor alternate reading frame protein (TARP) peptide vaccine: Will receive an admixture of the wildtype and epitope enhanced TARP peptides emulsified with Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF). TARP peptide will be administered subcutaneously at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.
- Arm B Autologous Dendritic Cell Vaccine: T-cell receptor alternate reading frame protein (TARP) dendritic cell vaccine: Will receive peptide pulsed dendritic cells administered intradermally in two vaccination sites. TARP pulsed dendritic cells will be administered at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.
Period: Overall Study
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Started | 21 | 20
Completed | 9 | 7
Not Completed | 12 | 13
Not completed — Switched to alternative treatment | 0 | 2
Not completed — Refused further treatment | 0 | 1
Not completed — Late determination of ineligibility | 0 | 1
Not completed — Second malignancy | 1 | 1
Not completed — Visa issues | 0 | 1
Not completed — Secondary cancer (SCC) | 0 | 1
Not completed — Met off study prostate specific antigen doubling time (PSADT) criteria | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Disease progression on study | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.58 (6.84) | 62.67 (7.4) | 63.14 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Baseline Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 3.44 [0.64 to 16.70] | 2.74 [0.48 to 30.70] | 3.44 [0.48 to 30.70]
Pre-Treatment Slope Log Prostate-Specific Antigen (PSA) [Median (Full Range); unit: Slope log] — "PSA slope log" calculated using Memorial Sloan Kettering Cancer Center Prostate Cancer Nomograms (http://nomograms.mskcc.org/Prostate/PsaDoublingTime.aspx) Slope log represents the speed of change of a series of values. Thus, it is reported without any units as it is with a concept of ratio which does not have any unit by its nature. The clinical meaning of PSA slope change would be decrease/increase of the "speed(velocity)" of changes in PSA, not the changes in PSA values. Decreasing PSA slope after the investigational treatment would mean the PSA rise is slower than pre-treatment baseline.
  Slope log | 0.087 [0.025 to 0.157] | 0.110 [0.054 to 0.239] | 0.101 [0.025 to 0.239]
Pre-Treatment Prostate-Specific Antigen Doubling Time (PSADT) [Median (Full Range); unit: Months] | 8.0 [4.4 to 27.7] | 6.3 [2.9 to 12.8] | 6.9 [2.9 to 27.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Immune Response Following Vaccination Determined by Interferon (IFN) Gamma Enzyme-linked Immunosorbent Spot (ELISpot)
Description: The number of participants in each arm with positive response determined by 3-fold increase over baseline in the number of positive cells by interferon (IFN) gamma enzyme-linked immunosorbent spot (ELISpot) at week 24. Presence of tumor antigen-specific T cells (positive response) mean the vaccine was able to generate immune response (i.e. immunogenicity) which is a good outcome.
Time Frame: Week 24
Population: 8/21 participants in Arm A and 4/20 participants in Arm B did not have samples available to analyze.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Number analyzed (Participants) | 13 | 16
Participants | 12 | 10

2. Primary Outcome: Grades 1-5 Adverse Events Possibly, Probably, or Definitely Related to Drug
Description: Adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: From date treatment consent signed and continuously through 30 days after last vaccination, approximately 59 months and 16 days for Arm A and 58 months and 24 days for Arm B.
Measure: Number; unit: Adverse Events
Groups:
- Arm B Autologous Dendritic Cell Vaccine: T-cell receptor alternate reading frame protein (TARP) peptide vaccine: Will receive an admixture of the wildtype and epitope enhanced TARP peptides emulsified with Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF). TARP peptide will be administered subcutaneously at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Number analyzed (Participants) | 21 | 20
Adverse Events
  Grade 1 Injection site reaction/extravasation changes definitely related to drug | 21 | 0
  Grade 2 Injection site reaction/extravasation changes definitely related to drug | 15 | 0
  No Grades 1-5 possibly and probably related to drug | 0 | 0
  No Grades 3-5 definitely related to drug | 0 | 0

3. Primary Outcome: Number of Participants With an Immunological Response of Chromium 51 (51Cr) Release Measured by Tetramer Staining OR Interferon (IFN)-Gamma Enzyme-linked Immune Absorbent Spot (ELISPOT) Assay
Description: A three-fold increase over baseline in the number of positive cells by tetramer staining OR Interferon (IFN)-gamma enzyme-linked immune absorbent spot (ELISPOT) assay was considered a positive immunological response.
Time Frame: Weeks 0, 12, 18 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Number analyzed (Participants) | 21 | 20
Participants
  Week 0 | 21 | 10
  Week 12 | 21 | 14
  Week 24 | 21 | 13

4. Secondary Outcome: PSA Doubling Time (PSADT) Response and Failure
Description: PSADT response is defined as: a > 50% increase in calculated PSADT OR a PSADT > 15 months. Participant's whose PSADT is decreased by > 50% will be considered PSADT failures. Week 24 PSADT responders will be allowed to receive an additional dose of T-cell receptor alternate reading frame protein (TARP) peptide vaccine at Week 36.
Time Frame: Weeks 12, 24, 36, and 48
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Number analyzed (Participants) | 21 | 20
Participants
  Week 12: ≥ 50% increase in calculated PSADT OR a PSADT > 15 months | 12 | 9
  Week 24: ≥ 50% increase in calculated PSADT OR a PSADT > 15 months | 13 | 11
  Week 36: ≥ 50% increase in calculated PSADT OR a PSADT > 15 months | 12 | 10
  Week 48: ≥ 50% increase in calculated PSADT OR a PSADT > 15 months | 9 | 10
  Week 12: PSADT is decreased by > 50% | 2 | 0
  Week 24: PSADT is decreased by > 50% | 0 | 0
  Week 36: PSADT is decreased by > 50% | 0 | 0
  Week 48: PSADT is decreased by > 50% | 0 | 0

5. Secondary Outcome: Change in Tumor Growth Rate Constant: Pre-versus Post T-cell Receptor Alternate Reading Frame Protein (TARP) Vaccination
Description: Changes in tumor growth rate constants (g) was calculated from fitting the prostate-specific antigen (PSA) curves to an exponential tumor growth model. Comparison of the median growth rate constant to 75th percentile [upper quartile]) of the estimated g of individual subjects pre- and post-TARP vaccination. The Tumor Growth Rate Constant was calculated using a regression-growth equation: f(t) = exp(-d x t) + exp(g x t) - 1, where exp is the base of the natural logarithm, e = 2.7182…, and f(t) is the PSA measurement at time t in days, normalized to (divided by) the PSA measurement at day 0, the time at which treatment is commenced. Rate constant d (decay, in days-1) represents the exponential decrease/regression rate constant of the PSA signal during therapy. Rate constant g (growth, also in days-1) represents the exponential growth/re-growth rate constant of the tumor during treatment.
Time Frame: 42-651 days on treatment
Population: Data was only available with participants combined for this outcome measure.
Measure: Number; unit: g = Days^(-1)
Groups:
- All Participants on Arm A and Arm B: Arm A Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF): T-cell receptor alternate reading frame protein (TARP) peptide vaccine: Will receive an admixture of the wildtype and epitope enhanced TARP peptides emulsified with Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF). TARP peptide will be administered subcutaneously at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.and Arm B Autologous Dendritic Cell Vaccine: T-cell receptor alternate reading frame protein (TARP) peptide vaccine: Will receive an admixture of the wildtype and epitope enhanced TARP peptides emulsified with Montanide ISA 51 VG and granulocyte-macrophage colony-stimulating factor (GM-CSF). TARP peptide will be administered subcutaneously at weeks 3, 6, 9, 12 and 15 for a total of five vaccinations with a booster dose of vaccine at Weeks 48 and 96.
Arm/Group | All Participants on Arm A and Arm B
Number analyzed (Participants) | 41
g = Days^(-1)
  Pre-vaccine | 0.0042
  Post-vaccine | 0.0021
Statistical Analysis 1: Comparison: All Participants on Arm A and Arm B; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
Number analyzed (Participants) | 21 | 20
Participants | 21 | 19

ADVERSE EVENTS:
Time Frame: From date treatment consent signed and continuously through 30 days after last vaccination, approximately 59 months and 16 days for Arm A and 58 months and 24 days for Arm B.
Arm/Group | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) | Arm B Autologous Dendritic Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/20
Other Adverse Events (participants affected / at risk) | 21/21 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) (N=21) | Arm B Autologous Dendritic Cell Vaccine (N=20)
Obstruction, Genitourinary: Ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain: Chest/Thorax Not Otherwise Specifed (NOS) (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Montanide ISA 51 VG and Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) (N=21) | Arm B Autologous Dendritic Cell Vaccine (N=20)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Denuded flaky area on the tip of penis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Dermatitis-like rash) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Cold sores) (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastrointestinal - Other (melena) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hemorrhage, gastrointestinal (GI)::Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Varices (rectal) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection - Other (Upper airway infection) (Infections and infestations) | 1 (2) | 0 (0)
Infection with normal absolute neutrophil count (ANC) or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Colon (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Eye NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 2 (2) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 21 (394) | 19 (190)
Insomnia (General disorders) | 1 (1) | 0 (0)
Leukocytes (total white blood cell (WBC) (Blood and lymphatic system disorders) | 2 (3) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5) | 7 (9)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/absolute granulocyte (AGC) (Blood and lymphatic system disorders) | 2 (3) | 1 (2)
Ocular/Visual - Other (Chalazion) (Eye disorders) | 1 (1) | 0 (0)
Pain - Other (Arthritis pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Abdomen NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (14) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0)
Vision-flashing lights/floaters (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT00972309/Prot_SAP_000.pdf
  • Informed Consent Form (2011-06-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT00972309/ICF_001.pdf